CLINICAL TRIAL: NCT01020903
Title: Aprepitant vs. Placebo for the Prevention of Postoperative Nausea and Vomiting: a Randomized, Double-blind Study in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Aprepitant for Post-operative Nausea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09-045
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Active Comparator)
  Interventions: Procedure: Aprepitant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Procedure: Aprepitant — 40 mg po pre-op
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — Orally, pre-op
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Anesthesia, especially for laparoscopic surgery, can cause post-operative nausea and vomiting. Most patients are given two drugs, decadron and ondansetron, to try to minimize this. This study is to determine if a new drug, aprepitant, would add any benefit in terms of post-op nausea prevention. All laparoscopic cholecystectomy study patients will receive decadron and ondansetron. Half the patients will receive aprepitant in addition. The other half will receive placebo. The study will be randomized and double-blind.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy patients.
* Must be able to swallow a pill.

Exclusion Criteria:

* Liver failure,
* Age less than 18.
* Pregnancy, breast-feeding.
* Pre-op vomiting.
* Allergy to aprepitant.
* Need for post-op gastric drainage.
* Use of drugs that interact with aprepitant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Silverberg, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

REFERENCES:
- [Background] Diemunsch P, Schoeffler P, Bryssine B, Cheli-Muller LE, Lees J, McQuade BA, Spraggs CF. Antiemetic activity of the NK1 receptor antagonist GR205171 in the treatment of established postoperative nausea and vomiting after major gynaecological surgery. Br J Anaesth. 1999 Feb;82(2):274-6. doi: 10.1093/bja/82.2.274. PMID 10365008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aprepitant | Placebo
Started | 100 (Please be advised that the investigator of the study left the institution in 2011.) | 100 (Please be advised that the investigator of the study left the institution in 2011.)
Completed | 100 (Please be advised that the investigator of the study left the institution in 2011.) | 100 (Please be advised that the investigator of the study entitled left the institution in 2011.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Records for this study are no longer available to the sponsor to update this study record as they were destroyed in Hurricane Sandy in 10/2012. thus, we do not have any information to use to update the records. PI for this study is no longer with the institution and no contact information is available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — Records for this study are no longer available to the sponsor to update this study record as they were destroyed in Hurricane Sandy in October 2012. This information was provided to FDA and OHRP when the event occurred in 2012. Thus, we do not have any information to use to update the records. In addition, the PI for this study is no longer with the institution and no contact information is available.
Sex/Gender, Customized [unit: participants]
Aprepitant vs Placebo [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Nausea and Vomiting
Description: Records for this study are no longer available to the sponsor to update this study record as they were destroyed in Hurricane Sandy in October 2012. This information was provided to FDA and OHRP when the event occurred in 2012. Thus, we do not have any information to use to update the records. In addition, the PI for this study is no longer with the institution and no contact information is available.
Time Frame: 1 year
Population: Records for this study are no longer available as they were destroyed in Hurricane Sandy in 10/2012- we do not have any information to use to update the records. The PI for this study is no longer with the institution and no contact information is available. Since we cannot verify the # of participants analyzed, the numbers were changed to "0".
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Aprepitant: Aprepitant: 40 mg po pre-op Please be advised that the investigator of the study entitled "Aprepitant for Post-operative Nausea" NCT01020903 left the institution in 2011. Normally, to update this record in clinicaltrial.gov, we would go to the IRB records. However, the IRB records of the reviewing IRB (Staten Island University Hospital IRB) were destroyed in Hurricane Sandy in October 2012. This information was provided to FDA and OHRP when the event occurred in 2012. Thus, we do not have any information to use to update the records.
- Placebo: Placebo: Orally, pre-op Please be advised that the investigator of the study entitled "Aprepitant for Post-operative Nausea" NCT01020903 left the institution in 2011. Normally, to update this record in clinicaltrial.gov, we would go to the IRB records. However, the IRB records of the reviewing IRB (Staten Island University Hospital IRB) were destroyed in Hurricane Sandy in October 2012. This information was provided to FDA and OHRP when the event occurred in 2012. Thus, we do not have any information to use to update the records.
Arm/Group | Aprepitant | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes